CLINICAL TRIAL: NCT05715528
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of GS-5245 for the Treatment of COVID-19 in Nonhospitalized Participants
Brief Title: Study of Obeldesivir in Nonhospitalized Participants With COVID-19
Acronym: OAKTREE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-611-6549; jRCT2031230285 (Other: Japan Registry of Clinical Trials)
Record Dates: First submitted 2023-02-03; First posted 2023-02-08 (Actual); Results first posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Participants, personnel directly involved in the conduct of study, and sponsor will not know the treatment participants received.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Obeldesivir (Experimental): Participants will receive obeldesivir 350 mg twice daily for 5 days.
  Interventions: Drug: Obeldesivir
- Obeldesivir Placebo (Placebo Comparator): Participants will receive obeldesivir placebo twice daily for 5 days.
  Interventions: Drug: Obeldesivir Placebo

INTERVENTIONS:
Drug: Obeldesivir — Tablet administered orally without regard to food.
  Other Names: GS-5245
  Arms: Obeldesivir
Drug: Obeldesivir Placebo — Tablet administered orally without regard to food.
  Arms: Obeldesivir Placebo

SUMMARY:
The goal of this clinical study is to test if obeldesivir (GS-5245) is safe and effective for the treatment of coronavirus disease 2019 (COVID-19) in participants who have a standard risk of developing severe illness. This study will also measure how much obeldesivir gets into the blood and how long it takes for the body to get rid of it.

ELIGIBILITY:
Key Inclusion Criteria:

* Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection confirmed, ≤ 3 days before randomization, by polymerase chain reaction (PCR), rapid antigen test, or an approved alternative assay. Serologic tests will not be accepted.
* Willing and able to complete the coronavirus disease 19 (COVID-19) symptom questionnaire prior to first dose and daily throughout the study period.
* Initial onset of COVID-19 signs/symptoms ≤ 3 days before randomization with ≥ 2 of the following targeted symptoms, at moderate or higher severity, present at randomization.

  * Stuffy or runny nose.
  * Sore throat.
  * Shortness of breath (difficulty breathing).
  * Cough.
  * Low energy or tiredness.
  * Muscle or body aches.
  * Headache.
  * Chills or shivering.
  * Feeling hot or feverish.
* Not currently hospitalized or requiring hospitalization.

Key Exclusion Criteria:

* Any risk factors for progression to severe disease.
* Planning to receive a direct acting antiviral or monoclonal antibody against SARS-CoV-2 for the treatment of COVID-19.
* Received any direct acting antiviral drug or monoclonal antibody against SARS-CoV-2 for the treatment of COVID-19 < 28 days or < 5 half-lives, whichever is longer, before randomization.
* Received any convalescent COVID-19 plasma or other antibody-based anti-SARS-CoV-2 prophylaxis at any time prior to study entry.
* Received an COVID-19 vaccine (including booster dose) < 120 days before randomization.
* Self-reported COVID-19 diagnosis < 120 days before randomization.
* Anticipated need for hospitalization < 48 hours after randomization.
* New oxygen requirement < 24 hours before randomization.
* Known influenza, or any other suspected or confirmed concurrent active systemic infection other than COVID-19 that may interfere with the evaluation of response to the study drug.
* Known history of chronic liver disease, limited to cirrhosis, nonalcoholic steatohepatitis, alcoholic liver disease, and autoimmune hepatitis.
* Undergoing dialysis, or known history of chronic kidney disease.
* Persistent symptoms from previous COVID-19 illness that may interfere with the evaluation of response to the study drug.
* Pregnant or breastfeeding.
* Unwilling to use protocol-mandated contraception.
* Any other factor, including inability to complete the patient-reported outcome (PRO) questionnaire for the primary endpoint, making the individual, in the opinion of the investigator, unsuitable to participate in the study.
* Concurrent participation/enrollment in a separate therapeutic clinical study.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 12 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2011 (Actual)
Dates: Start 2023-02-08 (Actual); Primary Completion 2023-11-28 (Actual); Study Completion 2024-01-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (112):
- United States (107):
  - EmVenio Research, Alabaster, Alabama
  - Institute for Liver Health dba Arizona Clinical Trials, Chandler, Arizona
  - The Institute for Liver Health dba Arizona Liver Health, Tucson, Arizona
  - Franco Felizarta, MD, Bakersfield, California
  - Velocity Clinical Research, Banning (IP Delivery and Administering Location), Banning, California
  - Benchmark Research, Colton, California
  - Ascada Research, Fullerton, California
  - Velocity Clinical Research, La Mesa, California
  - IMAX Clinical Trials, LLC, La Palma, California
  - Om Research LLC, Lancaster, California
  - L.A. Universal Research Center, INC., Los Angeles, California
  - Amicis Research Center, Northridge, California
  - Valley Clinical Trials, Northridge, California
  - Fomat Medical Research, Oxnard, California
  - Paradigm Clinical Research, Redding, California
  - Zuckerberg San Francisco General Hospital, San Francisco, California
  - Clearview Medical Research, LLC, Santa Clarita, California
  - EmVenio Research, Santa Monica, California
  - Med Partners, Inc. dba Premiere Medical Center of Burbank, Inc., Toluca Lake, California
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Encore Medical Research of Boynton Beach LLC, Boynton Beach, Florida
  - Palm Harbor Dermatology d/b/a TrueBlue Clinical Research, Brandon, Florida
  - Innovative Research of West Florida, Inc, Clearwater, Florida
  - Prestige Clinical Research Center Inc, Coral Gables, Florida
  - Beautiful Minds Clinical Research Center, Cutler Bay, Florida
  - Vital Care Research, Doral, Florida
  - UHC Research, LLC, Doral, Florida
  - Proactive Clinical Research,LLC, Fort Lauderdale, Florida
  - Qway Research LLC, Hialeah, Florida
  - AGA Clinical Trials, Hialeah, Florida
  - Research in Miami, Hialeah, Florida
  - 3Sync, LLC, Hialeah, Florida
  - Best Quality Research, Inc., Hialeah, Florida
  - Doral Medical Research, Hialeah, Florida
  - Evolution Clinical Trials, INC, Hialeah Gardens, Florida
  - Innovative Health, Hollywood, Florida
  - Encore Medical Research, LLC, Hollywood, Florida
  - Advance Clinical Research Group, Miami, Florida
  - Med-Care Research, Corp, Miami, Florida
  - Southern Clinical Research LLC, Miami, Florida
  - LCC Medical Research Institute, LLC, Miami, Florida
  - Universal Medical and Research Center, LLC., Miami, Florida
  - CCM Clinical Research Group, LLC, Miami, Florida
  - Global Health Clinical Trials Corp, Miami, Florida
  - Retreat Medical Research, Miami, Florida
  - Verus Clinical Research, Corp, Miami, Florida
  - Clinical Trial Services, Corp, Miami, Florida
  - Continental Clinical Research, Miami, Florida
  - Dynamic Medical Research, LLC, Miami, Florida
  - Nuren Medical & Research Center, Miami, Florida
  - Advanced Care and Clinical Trials, LLC, Miami, Florida
  - Bioclinical Research Alliance Inc., Miami, Florida
  - Cordova Research Institute, Inc, Miami, Florida
  - D&H National Research Centers, INC, Miami, Florida
  - Florida International Medical Research, Miami, Florida
  - Miami Clinical Research, Miami, Florida
  - Allied Biomedical Research Institute, Miami, Florida
  - Diverse Clinical Research, LLC, Miami, Florida
  - P&S Research, LLC., Miami, Florida
  - ProLive Medical Research, Corp, Miami, Florida
  - Entrust Clinical Research, Miami, Florida
  - Links Clinical Trials LLC, Miami, Florida
  - Reed Medical Research Corp, Miami, Florida
  - MedBio Trials LLC, Miami, Florida
  - Clinical Site Partners, LLC dba Flourish Research, Miami, Florida
  - Phoenix Research Center, LLC, Miami, Florida
  - Essential Clinical Research, Miami Lakes, Florida
  - Palm Springs Community Health Center, Miami Lakes, Florida
  - Angels Clinical Research Institute, Miami Lakes, Florida
  - Quality Research of South Florida, Miami Lakes, Florida
  - Oceanic Research Group, North Miami Beach, Florida
  - Castillo Torres, MD PA, Palm Springs, Florida
  - Family Clinical Trials, LLC, Pembroke Pines, Florida
  - USPA Advance Concept Medical Research Group, LLC, South Miami, Florida
  - Precision Clinical Research, Sunrise, Florida
  - Angels Clinical Research Institute, Tampa, Florida
  - Precision Research Center, Tampa, Florida
  - Santos Research Center, CORP, Tampa, Florida
  - Encore Medical Reseach of Weston, LLC, Weston, Florida
  - Clinical Site Partners, LLC dba Flourish Research, Winter Park, Florida
  - EmVenio Research, Atlanta, Georgia
  - Agile Clinical Research Trials, LLC, Atlanta, Georgia
  - Covenant Pulmonary Critical Care Research Institute, East Point, Georgia
  - Velocity Clinical Research, Lafayette, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Prime Global Research Inc, The Bronx, New York
  - Shelby Clinical Research, LLC, Denver, North Carolina
  - The Brody School of Medicine at East Carolina University, Greenville, North Carolina
  - Carolina Research Center, Inc., Shelby, North Carolina
  - Frontier Clinical Research, LLC, Smithfield, Pennsylvania
  - Clinovacare Medical Research Center, West Columbia, South Carolina
  - St Hope Foundation, Inc., Bellaire, Texas
  - PanAmerican Clinical Research, Brownsville, Texas
  - Premier Pulmonary Critical Care and Sleep Medicine, Denison, Texas
  - EmVenio Research, Fort Worth, Texas
  - HDH Research Inc., Houston, Texas
  - The Crofoot Research Center, INC., Houston, Texas
  - Milton Haber, MD, Laredo, Texas
  - SMS Clinical Research, LLC, Mesquite, Texas
  - Village Health Partners, Plano, Texas
  - North Texas Family Medicine, Plano, Texas
  - Epic Medical Research, LLC, Red Oak, Texas
  - STAAMP Research LLC, San Antonio, Texas
  - Tranquil Clinical Research, Webster, Texas
  - Bountiful Internal Medicine, Bountiful, Utah
  - Velocity Clinical Research, Salt Lake City, West Jordan, Utah
  - Frontier Clinical Research, LLC, Kingwood, West Virginia
- Japan (5):
  - Kanagawa Himawari Clinic, Kawasaki-Shi
  - Medical corporation Shirayurikai Swing Nozaki Clinic, Musashino
  - Nishioka Hospital, Sapporo-Shi Toyohira-Ku
  - Sato Clinic, Shibuya-ku
  - Tokyo Shinagawa Hospital Social Medical Corporation Association Tokyokyojuno-kai, Shinagawa-Ku

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rodriguez L, Hu Y, Li J, Han D, Peinovich N, Martinez C, Ho PY, Perry JK, Martin R, Ogbuagu O, Lichtman A, Hyland RH, Hedskog C. SARS-CoV-2 Resistance Analyses From the Phase 3 OAKTREE Study of Obeldesivir in Low-Risk Nonhospitalized Participants With COVID-19. Antiviral Res. 2025 Dec 29:106339. doi: 10.1016/j.antiviral.2025.106339. Online ahead of print. PMID 41475511
- [Derived] Ogbuagu O, Goldman JD, Gottlieb RL, Singh U, Shinkai M, Acloque G, Fusco DN, Gonzalez E, Kumar P, Luetkemeyer A, Lichtman A, Mozaffarian A, Koullias Y, Hyland RH, Llewellyn J, Osinusi A, Duff F, Humeniuk R, Caro L, Davies S, Rodriguez L, Hedskog C, Chen S, Etchevers K, Nadig P, Kohli A; OAKTREE Trial Investigators. Efficacy and safety of obeldesivir in low-risk, non-hospitalised patients with COVID-19 (OAKTREE): a phase 3, randomised, double-blind, placebo-controlled study. Lancet Infect Dis. 2025 Dec;25(12):1282-1292. doi: 10.1016/S1473-3099(25)00238-5. Epub 2025 Jul 14. PMID 40675167
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=GS-US-611-6549

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 2253 participants were screened.
Pre-assignment Details: Participants were enrolled at study sites in the United States and Japan.
Groups:
- Obeldesivir: Participants received obeldesivir 350 mg orally twice daily without regard to food for 5 days.
- Placebo: Participants received placebo-to-match obeldesivir orally twice daily without regard to food for 5 days.
Period: Overall Study
Arm/Group | Obeldesivir | Placebo
Started | 1005 | 1006
Completed | 977 | 963
Not Completed | 28 | 43
Not completed — Randomized but never treated | 11 | 13
Not completed — Withdrew consent | 7 | 15
Not completed — Lost to Follow-up | 5 | 13
Not completed — Investigator's discretion | 3 | 1
Not completed — Protocol Violation | 2 | 0
Not completed — Non-compliance with study drug | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all participants, who were randomized into the study and have received at least 1 dose of study drug, except from one of the site which did not comply with study rules.
Groups:
- Total: Total of all reporting groups
Arm/Group | Obeldesivir | Placebo | Total
Number analyzed (Participants) | 979 | 976 | 1955
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 19 | 15 | 34
  Between 18 and 65 years | 960 | 961 | 1921
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (12.9) | 41 (12.3) | 41 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 583 | 572 | 1155
  Male | 396 | 404 | 800
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 918 | 901 | 1819
  Not Hispanic or Latino | 61 | 75 | 136
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 3 | 3
  Asian | 21 | 21 | 42
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 106 | 101 | 207
  White | 850 | 848 | 1698
  More than one race | 1 | 3 | 4
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 962 | 962 | 1924
  Japan | 17 | 14 | 31
Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) viral load [Mean (Standard Deviation); unit: log10 copies/mL] | 5.08 (1.416) | 5.09 (1.479) | 5.09 (1.448)

OUTCOME MEASURES:

1. Primary Outcome: Time to Coronavirus Disease 2019 (COVID-19) Symptom Alleviation by Day 29
Description: The time to alleviation of targeted COVID-19 symptoms by Day 29 for participants with symptom alleviation, was calculated as symptom alleviation date/time minus first dose date/time. For participants who completed Day 29 of the study or discontinued from the study before Day 29 without symptom alleviation (censored) and without inter-current events, time was calculated as last date/time on which symptom alleviation was assessed minus the first dose date/time or Day 28, whichever occurred first. Symptom alleviation was defined as, all targeted symptoms scored moderate or severe at baseline were scored as mild/none and all targeted symptoms scored mild/none at baseline were scored as none, for at least 48 consecutive hours. Targeted symptoms included: stuffy or runny nose, sore throat, shortness of breath, cough, low energy or tiredness, muscle or body aches, headache, chills or shivering and feeling hot or feverish.
  Kaplan-Meier (KM) estimates were used in outcome measure analysis.
Time Frame: First dose date up to Day 29
Population: The Full Analysis Positive Set (FAPS) included all participants, except from one of the site which did not comply with study rules, who were randomized into the study, have received at least 1 dose of study drug, and were SARS-CoV-2 positive at baseline as confirmed by Cepheid's Xpert Xpress CoV-2/Flu/RSV plus test or SARS-CoV-2 reverse transcriptase-quantitative polymerase chain reaction (RT-qPCR) test from central lab.
  Participants with available data were analyzed.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Obeldesivir | Placebo
Number analyzed (Participants) | 879 | 882
days | 5.9 [5.4 to 6.1] | 6.0 [5.8 to 6.3]
Statistical Analysis 1: Comparison: Obeldesivir vs Placebo; Test type: Superiority; p = 0.0681, Stratified Log-rank test — P-value calculated from stratified Log-rank test with randomization stratification factor as the strata; Hazard Ratio (HR) = 1.099, 95% CI 2-sided [0.997 to 1.211] — Hazard ratio and two-sided 95% confidence interval (CI) for hazard ratio were estimated using the Cox regression with randomization stratification factor as a covariate

2. Primary Outcome: Percentage of Participants Experiencing Treatment-emergent Adverse Events (TEAEs)
Description: TEAEs were defined as 1 or both of the following:
  * Any AEs with an onset date on or after the study drug start date and no later than 30 days after permanent discontinuation of study drug.
  * Any AEs leading to premature discontinuation of study drug. Percentages were rounded off.
Time Frame: First dose date up to Day 5 plus 30 days
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Obeldesivir | Placebo
Number analyzed (Participants) | 979 | 976
percentage of participants | 5.4 | 5.7

3. Primary Outcome: Percentage of Participants Experiencing Laboratory Abnormalities
Description: Treatment-emergent laboratory abnormalities were defined as values that increase at least 1 toxicity grade from baseline at any postbaseline time point, up to and including the date of last dose of study drug plus 30 days.
  Percentages were rounded off.
Time Frame: First dose date up to Day 5 plus 30 days
Population: Participants from the Safety Analysis Set who had available postbaseline data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Obeldesivir | Placebo
Number analyzed (Participants) | 972 | 964
percentage of participants
  Any grade | 77.5 | 78.5
  Grade 3 or 4 | 6.1 | 8.5

4. Primary Outcome: Percentage of Participants Experiencing Serious Adverse Events (SAEs) and Adverse Events (AEs) Leading to Study Drug Discontinuation
Description: Percentages were rounded off.
Time Frame: First dose date up to Day 5 plus 30 days
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Obeldesivir | Placebo
Number analyzed (Participants) | 979 | 976
percentage of participants
  SAEs | 0.2 | 0.4
  AEs leading to study drug discontinuation | 0.1 | 0

5. Secondary Outcome: Time to COVID-19 Symptom Resolution by Day 29
Description: COVID-19 symptom resolution was defined as all targeted symptoms scored as none for at least 48 consecutive hours. The first day of the 48 consecutive hours was considered the date of symptom resolution. The time to COVID-19 symptom resolution was the time (expressed as days) from the first dose date/time to the date/time of symptom resolution.
  KM estimates were used in the outcome measure analysis.
Time Frame: Day 1 up to 29
Population: Participants in the Full Analysis Positive Set with available data were analyzed.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Obeldesivir | Placebo
Number analyzed (Participants) | 879 | 882
days | 9.2 [8.9 to 10.0] | 9.3 [8.9 to 10.1]
Statistical Analysis 1: Comparison: Obeldesivir vs Placebo; Test type: Superiority; p = 0.5558, Stratified Log-Rank Test; P-value calculated from stratified Log-rank test with randomization stratification factor as the strata; Hazard Ratio (HR) = 1.036, 95% CI 2-sided [0.935 to 1.147] — Hazard ratio and two-sided 95% CI for hazard ratio were estimated using the Cox regression with randomization stratification factor as a covariate

6. Secondary Outcome: Percentage of Participants With Moderate Relapse of COVID-19 Symptoms by Day 29
Description: COVID-19 moderate symptom relapse was defined as having at least 1 symptom being moderate or severe OR at least 2 mild symptoms OR a hospitalization for COVID-19 or death, observed on a day during COVID-19 symptom relapse.
  Percentages were rounded off.
Time Frame: Up to Day 29
Population: Participants in the Full Analysis Positive Set who had short symptom recovery with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Obeldesivir | Placebo
Number analyzed (Participants) | 760 | 743
percentage of participants | 8.3 [6.4 to 10.5] | 9.0 [7.1 to 11.3]
Statistical Analysis 1: Comparison: Obeldesivir vs Placebo; Test type: Superiority; p = 0.6469, Fisher's exact test

7. Secondary Outcome: Percentage of Participants With COVID-19 Related Medically Attended Visits (MAVs) or All-cause Death by Day 29
Description: Medically attended visits were defined as interactions with health care professionals other than study staff or designees including hospitalization; in-person emergency, urgent, or primary care visits; or any other in-person visit attended by the participant and a health care professional. The nature and cause of the visit were identified.
  KM estimates were used in the outcome measure analysis. Percentages were rounded off.
Time Frame: Up to Day 29
Population: Participants in the Full Analysis Positive Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Obeldesivir | Placebo
Number analyzed (Participants) | 884 | 884
percentage of participants | 0.1 [0.0 to 0.3] | 0.2 [0.0 to 0.5]
Statistical Analysis 1: Comparison: Obeldesivir vs Placebo; Test type: Superiority; p = 0.5581, Log-rank test; P value was based on log-rank test; Hazard Ratio (HR) = 0.495, 95% CI 2-sided [0.045 to 5.464] — Hazard ratio and two-sided 95% CI were estimated using the Cox regression

8. Secondary Outcome: Percentage of Participants With COVID-19 Related Hospitalization or All-cause Death by Day 29
Description: COVID-19-related hospitalization was defined as ≥ 24 hours of acute care for a reason related to COVID-19, in a hospital or similar acute care facility, including emergency rooms or temporary facilities instituted to address medical needs of those with COVID-19. This included specialized acute medical care units within an assisted living facility or nursing home. This did not include hospitalization for the purposes of public health and/or clinical trial execution. The date and duration (if there was 1 day difference between the start date and end date) of hospital admission, and primary reason for hospitalization (including if the hospitalization was related to COVID-19) was to be recorded.
  Percentages were rounded off.
Time Frame: Up to Day 29
Population: Participants in the Full Analysis Positive Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Obeldesivir | Placebo
Number analyzed (Participants) | 884 | 884
percentage of participants | 0 | 0

9. Secondary Outcome: Change From Baseline in Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) Nasal Swab Viral Load at Day 5
Time Frame: Day 5
Population: The Virology Analysis Set included all participants, who were randomized into the study, had received at least 1 dose of study drug, and had a baseline SARS-CoV-2 viral load ≥ Lower limit of quantification (LLOQ).
  Participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: log10 copies/mL
Arm/Group | Obeldesivir | Placebo
Number analyzed (Participants) | 637 | 622
log10 copies/mL | -2.69 (0.019) | -2.71 (0.020)
Statistical Analysis 1: Comparison: Obeldesivir vs Placebo; Test type: Superiority; p = 0.4254, MMRM — p-value was from Mixed-effects model repeated measures (MMRM) with baseline viral load and randomization strata as covariates; Least Squares Mean = 0.02, 95% CI 2-sided [-0.03 to 0.08] — 95% CI was from MMRM with baseline viral load and randomization strata as covariates

10. Secondary Outcome: Time to Antigen Negativity
Description: Time to antigen negativity was defined (in days) as the number of days to the first date of 2 consecutive dates achieving a negative result. Antigen negativity was defined as 2 consecutive negative SARS-CoV-2 rapid antigen test (regardless if there was missing data in between), or negative test at last available sample for participants who completed or discontinued from the study after at least 1 positive antigen test.
Time Frame: Day 1 up to Day 29
Population: The Antigen Analysis Set included all participants, who were randomized into the study, had received at least 1 dose of study drug, and had at least 1 SARS-CoV-2 rapid antigen test positive from Day 1 to Day 5 and SARS-CoV-2 polymerase chain reaction (PCR) positive at baseline per Full Analysis Positive Set.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Obeldesivir | Placebo
Number analyzed (Participants) | 809 | 803
days | 5.0 [3.0 to 6.0] | 5.0 [4.0 to 6.0]
Statistical Analysis 1: Comparison: Obeldesivir vs Placebo; Test type: Superiority; p = 0.0015, Stratified Log-rank test — P-value calculated from stratified Log-rank test with randomization stratification factor as the strata; Hazard Ratio (HR) = 1.138, 95% CI 2-sided [1.032 to 1.256] — [estimate comment as in outcome 5, analysis 1]

11. Secondary Outcome: Percentage of Participants With Viral Antigen Rebound
Description: Viral antigen rebound was defined as any positive SARS-CoV-2 rapid antigen test after antigen negativity.
  Percentages were rounded off.
Time Frame: Up to Day 29
Population: Participants from Antigen Analysis Set with antigen negativity were included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Obeldesivir | Placebo
Number analyzed (Participants) | 809 | 803
percentage of participants | 1.5 [0.8 to 2.6] | 1.7 [1.0 to 2.9]
Statistical Analysis 1: Comparison: Obeldesivir vs Placebo; Test type: Superiority; p = 0.6978, Fisher's exact test; P-value was from the Fisher's exact test

12. Secondary Outcome: Plasma Concentrations of GS-441524 (Metabolite of Obeldesivir)
Time Frame: Day 1, 0.75 hour and 2 hours; Day 3, Predose and 0.75 hour; Day 5, Predose and 0.75 hour
Population: The Pharmacokinetic (PK) Analysis Set included all randomized participants, who took at least 1 dose of study drug and had at least 1 non-missing concentration value reported by the PK laboratory for GS-441524.
  Participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Obeldesivir
Number analyzed (Participants) | 940
ng/mL
  Day 1 (0.75 h): number analyzed (Participants) | 831
  Day 1 (0.75 h) | 2528.97 (5633.223)
  Day 1 (2 h): number analyzed (Participants) | 709
  Day 1 (2 h) | 2390.68 (4763.877)
  Day 3 (Predose): number analyzed (Participants) | 887
  Day 3 (Predose) | 1103.79 (6500.997)
  Day 3 (0.75 h): number analyzed (Participants) | 655
  Day 3 (0.75 h) | 3339.59 (11353.578)
  Day 5 (Predose): number analyzed (Participants) | 661
  Day 5 (Predose) | 2599.61 (29678.065)
  Day 5 (0.75 h): number analyzed (Participants) | 570
  Day 5 (0.75 h) | 4595.37 (30772.089)

13. Secondary Outcome: Pharmacokinetic (PK) Parameter: AUCtau,Steady-State of GS-441524
Description: AUCtau is defined as the area under the concentration versus time curve over the dosing interval at steady-state.
Time Frame: Day 5
Population: The Intensive PK Substudy analysis set included all randomized participants, who took at least 1 dose of study drug, participated in the intensive PK substudy, and had at least 1 non-missing concentration for GS-441524, excluding participants with identified outliers, were analyzed.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Obeldesivir
Number analyzed (Participants) | 63
h*ng/mL | 18000 (10200)

14. Secondary Outcome: PK Parameter: Ctau of GS-441524
Description: Ctau is defined as the observed drug concentration at the end of the dosing interval.
Time Frame: Day 1 and Day 5
Population: Participants from Intensive PK Substudy Analysis Set excluding participants with identified outliers, were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Obeldesivir
Number analyzed (Participants) | 64
ng/mL
  Day 1: number analyzed (Participants) | 54
  Day 1 | 772 (761)
  Day 5 | 735 (919)

15. Secondary Outcome: PK Parameter: Cmax of GS-441524
Description: Cmax is defined as the maximum observed plasma concentration of drug.
Time Frame: Day 1 and Day 5
Population: Participants from Intensive PK Substudy Analysis Set excluding participants with identified outliers, were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Obeldesivir
Number analyzed (Participants) | 99
ng/mL
  Day 1 | 2910 (1010)
  Day 5: number analyzed (Participants) | 68
  Day 5 | 2920 (1220)

16. Secondary Outcome: Percentage of Participants With Relapse of COVID-19 Symptoms by Day 29
Description: Symptom relapse means at least 2 consecutive diary entries (regardless of missing data in between) where there was any symptom (regardless of severity) OR a hospitalization for COVID-19 or a death after short symptom recovery.
  Percentages were rounded off.
Time Frame: Up to Day 29
Population: Participants in the Full Analysis Positive Set with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Obeldesivir | Placebo
Number analyzed (Participants) | 760 | 743
percentage of participants | 10.9 [8.8 to 13.4] | 12.0 [9.7 to 14.5]
Statistical Analysis 1: Comparison: Obeldesivir vs Placebo; Test type: Superiority; p = 0.5707, Fisher's exact test; P-value was from the Fisher's exact test

ADVERSE EVENTS:
Time Frame: Adverse Events and All-Cause Mortality: Up to 35 days
Description: All-cause mortality: All Randomized Analysis Set included all participants who were randomized in the study.
  Adverse events: The Safety Analysis Set included all participants, who were randomized into the study and have received at least 1 dose of study drug, except from one of the site which did not comply with study rules.
Arm/Group | Obeldesivir | Placebo
All-Cause Mortality (participants affected / at risk) | 0/1005 | 0/1006
Serious Adverse Events (participants affected / at risk) | 2/979 | 4/976
Other Adverse Events (participants affected / at risk) | 0/979 | 0/976
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Obeldesivir (N=979) | Placebo (N=976)
Gastroenteritis bacterial (Infections and infestations) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Bipolar disorder (Psychiatric disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2023-12-12): https://cdn.clinicaltrials.gov/large-docs/28/NCT05715528/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-11): https://cdn.clinicaltrials.gov/large-docs/28/NCT05715528/SAP_001.pdf